CLINICAL TRIAL: NCT06397911
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Pharmacokinetics, and Safety of Repeat Subcutaneous Doses of FB825 in Adults With Moderate-to-Severe Atopic Dermatitis
Brief Title: Evaluate Efficacy and Safety of Repeat Subcutaneous Doses of FB825 in Adults With Moderate-to-Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB825CLRS02
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Biological: FB825 Other: Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FB825 (Experimental)
  Interventions: Drug: FB825
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB825 — The study treatment will be administered as 5 SC doses in total 12 weeks
  Arms: FB825
Drug: Placebo — The study treatment will be administered as 5 SC doses in total 12 weeks
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled and double-blind study to evaluate the efficacy, pharmacokinetics, and Safety of repeat subcutaneous doses of FB825 in adults with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled, 2-arm, parallel-group study will enroll approximately 90 subjects with moderate-to-severe atopic dermatitis, with approximately 45 subjects per group.

The study duration of subject participation in the study is up to 28 weeks, including up to 4 weeks for screening, a 12-week study intervention and a 12-week follow-up period after study intervention. The study treatment will be administered as 5 SC doses.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. The subject is male or female between 18 and 65 years of age at the time of giving informed consent.
2. Body weight equal to or greater than 40 Kg at the time of screening.
3. The subject has a physician-confirmed diagnosis of moderate-to-severe atopic dermatitis based on 12 months history of symptoms designated by Hanifin and Rajka criteria.
4. Eczema Area and Severity Index (EASI) score ≥16 at screening and baseline visits.
5. Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score ≥ 3 (5-point scale) at the screening and baseline visits.
6. ≥10 % body surface area (BSA) of AD involvement at the screening and baseline visits.
7. Baseline pruritus numerical rating scale (NRS) average score for maximum itch intensity of ≥ 3, based on the average of daily pruritus NRS scores for maximum itch intensity reported during the 7 days prior to randomization.
8. History of inadequate response to a stable (4 weeks) regimen of topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) as treatment for AD within 6 months before the screening visit. (The TCS should belong to medium to high potency strength and has been applied for at least 4 weeks or for the maximum duration recommended by product prescribing information.)

   * An inadequate response is defined as the inability to achieve and maintain remission or a low disease activity state (comparable to vIGA-AD 0=clear to 2=mild).
   * Subjects with systemic treatment for AD in the past 6 months were also considered as inadequate responders to topical treatments.
9. Patients must be applying stable doses of an additive-free, basic bland emollient twice-daily for at least 1 week immediately before the baseline visit.

   Note: See exclusion criterion #13 for limitations regarding emollients.
10. Female subjects must have a negative serum pregnancy test at screening. All subjects of childbearing potential and his/her sexual partner must meet 2 following condition or acceptable methods of birth control throughout the study.

    * Oral, injectable, or implanted hormonal contraceptives
    * Condom with a spermicidal form, gel, film, cream, or suppository
    * Occlusive cap (diaphragm or cervical/vault caps) with a spermicidal foam, gel, film, cream, or suppository
    * Intrauterine device
    * Intrauterine system (for example, progestin-releasing coil) or be surgically sterile (i.e., hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or vasectomy)
    * Postmenopausal (defined as amenorrhea 12 consecutive months and documented serum follicle stimulating hormone level per laboratory standard) Note: The subject must utilize the method of effective contraception during study period as well as 16 weeks or 5 half-lives following the last dosing of FB825.
11. The subject is able to provide written informed consent.
12. The subject agrees to and is capable of adhering to scheduled visits, the treatment plan, laboratory tests, other study procedures, and all protocol requirements.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Female subjects who are pregnant or lactating
  2. The subject with positive test results for HBeAg or HCV RNA should be excluded as they are indications of active hepatitis B virus and hepatitis C virus replication.
  3. A positive human immunodeficiency virus (HIV) test (e.g., HIV Ag/Ab combo test) at screening or a history of HIV infection.
  4. The subject has a history of alcohol or drug abuse within one year prior to screening that would impair or risk the patients' full participation in the study, in the opinion of the investigator.
  5. The subject has a clinically significant, currently active or severe gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory (with the exception of uncomplicated allergic rhinitis and allergic asthma), inflammatory, immunological, endocrine, diabetes, obesity [BMI≥35] or infectious disease and is ineligible to participate in the study as judged by the investigator.
  6. The subject has a clinically significant history, as determined by the investigator, of drug allergies or hypersensitivity such as, but not limited to, sulfonamides and penicillin, or a drug allergy witnessed in a previous study with experimental drugs.
  7. The subject has any history of a previous anaphylactic reaction.
  8. The subject has any condition that, in the opinion of the investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements.
  9. The subject has received TCS or TCI within 7 days prior to the baseline visit (Day 1).
  10. The subject has received any immunoglobulin products or blood products within 3 months prior to baseline visit.
  11. The subject has received a biologic product (including investigational biologic product) within 5 half-lives or 3 months, whichever is longer, before baseline visit.
  12. The subject has received an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before baseline visit.
  13. Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period.
  14. Initiation of treatment of AD with sedative anti-histamine products during the screening period (patients may continue using stable doses of non-sedative anti-histamine).
  15. The subject is a member of the professional or ancillary personnel involved in the study.
  16. The subject regular use (≥2 visits per week) of a tanning booth/parlor within 4 weeks prior to the baseline visit.
  17. The subject has received cell-based immunotherapy treatment within 3 months prior to baseline visit.
  18. The subject has used any of the following classes of medication (prescription or over-the-counter) within specific time frames before the study drug treatment:

      * Systemic corticosteroids within 4 weeks.
      * Leukotriene modifiers within 4 weeks.
      * Cyclosporine within 4 weeks, or other immunosuppressants (e.g. gold salts, methotrexate, azathioprine) within 4 weeks.
      * IFN-γ within 12 weeks, or other immunomodulating drugs within 4 weeks.
      * Allergen immunotherapy within 1 year.
      * JAK inhibitor within 4 weeks.
  19. The subject has received phototherapy within 4 weeks before the study drug treatment.
  20. The subject has received live vaccine within 12 weeks before the study drug treatment.
  21. The subject has presence of skin comorbidities that may interfere with study assessments.
  22. The subject has known or suspected history of immunosuppression, including history of opportunistic infections (e.g., TB) per investigator's judgment.
  23. The subject has active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit.

      Note: Patients with resolved infection may be rescreened.
  24. The subject has history of malignancy within 5 years before the screening period, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
  25. The subject has planned or anticipated the use of any prohibited medications and procedures during the entire study period.
  26. The subject has planned or anticipated major surgical procedure during the entire study period.
  27. High risk of parasite infection. Evidence of parasitic infection designated as having the following two items:

      • Risk factors for parasitic disease include living in an endemic area, experiencing chronic gastrointestinal symptoms, traveling to regions where geohelminthic infections are endemic within the last 6 months, and/or having chronic immunosuppression).

      AND

      • Evidence of parasitic colonization or infection found during stool evaluation for ova and parasites.

      Note: stool ova and parasite evaluation will only be conducted in patients with risk factors and an eosinophil count more than twice the upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change from baseline in Eczema Area and Severity Index (EASI) score | Week 16

SECONDARY OUTCOMES:
The percentage change from baseline in Eczema Area and Severity Index (EASI) score | Week 2, 4, 8, 12, 20 and 24
The mean change from baseline in Eczema Area and Severity Index (EASI) score | Week 2, 4, 8, 12, 16, 20, and 24
Proportion of patients with EASI-75 (≥75% improvement from baseline) | Week 2, 4, 8, 12, 16, 20, and 24
Proportion of patients with EASI-50 (≥50% improvement from baseline) | Week 2, 4, 8, 12, 16, 20, and 24
Proportion of patients with EASI-90 | Week 2, 4, 8, 12, 16, 20, and 24
The percentage change from baseline in Investigator Global Assessment (IGA) score | Week 2, 4, 8, 12, 16, 20, and 24
Proportion of patients with both Investigator Global Assessment (IGA) 0 to 1 and a reduction from baseline of ≥2 points | Week 2, 4, 8, 12, 16, 20, and 24
The percentage change from baseline in Severity Scoring of Atopic Dermatitis Index (SCORAD) score | Week 2, 4, 8, 12, 16, 20, and 24
The percentage change from baseline in pruritus numerical rating scale (NRS) score | Week 2, 4, 8, 12, 16, 20, and 24
The mean change from baseline in Dermatology Life Quality Index (DLQI) score | Week 2, 4, 8, 12, 16, 20, and 24
The percentage change from baseline in total IgE | Week 2, 4, 8, 12, 16, 20, and 24
The percentage change from baseline in allergen-specific IgE | Week 4, 16, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, Principal Investigator — National Taiwan University Hospital
Locations (16):
- United States (6):
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - University of California, Davis Health, Department of Dermatology, Sacramento, California
  - UT Health Science Houston, Bellaire, Texas
  - Center for Clinical Studies, Webster, Texas
- Taiwan (10):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Linkou Chang Gung Memorial Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei